CLINICAL TRIAL: NCT02857114
Title: Measuring the Effects of Touch Relaxation Painful Patients in Oncologie Nursing
Acronym: ToucherDétente
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014-20
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- massage (Other)
  Interventions: Other: massage

INTERVENTIONS:
Other: massage

SUMMARY:
Measure the impact of touch relaxation on pain communicative patients suffering from chronic pain of cancer origin inpatient Oncology. measure over three days the effects on pain anxiety welfare and consumption of analgesics

ELIGIBILITY:
Inclusion Criteria:

hospitalized in the oncology department at least 3 days

* presenting the cancerous type of pain caused by their disease or treatment
* numerical scale pain score = 4/10
* receiving weak and strong opioids
* platelet count> 100
* can receive anxiolytic
* adult
* Patient of both sexes
* no other relaxation approaches

Exclusion Criteria:

* against indication to touch: wound, bruises, circulatory disorders, diseases psychiatiques
* risk of hematoma
* numerical scale pain score < 4/10
* understanding of the difficulties of the French language
* no receiving weak and strong opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 3 days
  pain measurement by the scale numerical pain

SECONDARY OUTCOMES:
anxiety | 3 days
  measurement with the scale of COVI
consumption of analgesics | 3 days
  daily creel analgesics and anxiolytics
wellness | 3 days
  measure with the scale of edmonton

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France